CLINICAL TRIAL: NCT01092689
Title: Understanding the Role of Meat-Borne Carcinogen in Pancreatic Cancer Etiology
Brief Title: The Role of Meat-borne Carcinogens in Pancreatic Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Needed New IND per FDA
Sponsor: University of Minnesota (Other)
Collaborators: University of Arkansas (Other); Lawrence Livermore National Laboratory (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2007NT128
Record Dates: First submitted 2010-03-23; First posted 2010-03-25 (Estimated); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Pancreas Cancer
Keywords: heterocyclic amines; PhIP; Meat; pancreas neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 2-amino-1-methyl-6-phenylimidazo(4,5-b)pyridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PhIP (Experimental): Prior to surgery, consented subjects will ingest a capsule containing [14C]PhIP. This amount of [14C]PhIP (84 micrograms PhIP; 15.6 micro-curies) is equivalent to that in 2 very well done grilled/barbecued chicken breasts (Sinha 1995); the amount of radioactivity is equivalent to the dose received in a commercial airline flying at 30,000 ft. for 5 h (HPS 2007) or to the amount received during a typical chest x-ray.
  Interventions: Drug: PhiP

INTERVENTIONS:
Drug: PhiP — 1 capsule of 84 micrograms; 15.6 micro-curies [14C]PhIP

SUMMARY:
We propose to recruit subjects scheduled for pancreatectomy as a treatment for pancreatic cancer. These subjects will ingest a very low dose of radiolabeled PhIP, a meat-derived carcinogen, and a small amount of resected tissue (waste) will be analyzed with highly sensitive technology to determine if this carcinogen binds to DNA in the pancreas.

DETAILED DESCRIPTION:
Pancreatic cancer is rapidly fatal in most cases and little is known about its causes. Identifying and modifying risk factors can reduce mortality through prevention. Carcinogens that form in meat cooked at high temperatures may be modifiable risk factors for pancreatic cancer, but direct evidence is needed to demonstrate involvement in pancreas tissue. We propose to recruit subjects scheduled for pancreatectomy as a treatment for pancreatic cancer. These subjects will ingest a very low dose of radiolabeled PhIP, a meat-derived carcinogen, and a small amount of resected tissue (waste) will be analyzed with highly sensitive technology to determine if this carcinogen binds to DNA in the pancreas. We hypothesize that the meat-derived carcinogen will bind to DNA in the pancreas. The amount of PhIP ingested is equivalent to the amount in two very well-done barbecued chicken breasts and the dose of radioactivity is comparable to a typical chest x-ray. This research can increase understanding of pancreatic carcinogenesis, facilitating the design of prevention strategies.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old.
* Adequate hepatic function within 4 weeks of study enrollment defined as bilirubin ≤ 2 mg/dl and ALT, AST, and alkaline phosphatase ≤ 2 times the upper limit of normal.
* Females of childbearing potential or males whose partners are of child bearing potential are required to use an effective method of contraception (i.e., a hormonal contraceptive. intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) during the study and for 4 months after PhIP administration.
* Voluntary written informed consent (PhIP consent and Caffeine assay consent) before performance of any study-related procedure not part of normal medical care, with the understanding that the subject may withdraw consent at any time without prejudice to future medical care.

Exclusion Criteria:

* CA-19-9 equal to or above 400.
* Tumor size >3.5 cm.
* Fluid in the abdomen (ascites).
* Conditions present, which, in the opinion of the surgeon, could make resection difficult, e.g., extensive vascular involvement.
* Pregnant or lactating (for women).
* Uncontrolled cardiovascular disease; e.g. hypertension, angina, etc.
* Patients who are intolerant of a 200 mg dose of caffeine or who otherwise do not wish to participate in the caffeine assay when consent is sought for the primary consent will be considered refusers and will not be enrolled in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Quantify and characterize HCA-DNA adducts in resected human pancreatic tissue after a dietary relevant dose of PhIP, the most mass abundant HCA in charred meat. | 6 hours post ingestion

SECONDARY OUTCOMES:
Quantify [14C]PhIP and [14C]PhIP metabolites in urine and plasma. | From 0 to 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Kristin E Anderson, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States